CLINICAL TRIAL: NCT07317479
Title: Clinical Study for P-MAR Metal Artifact Reduction Algorithm for Incisive CT and CT 5300 Systems
Brief Title: Clinical Study for P-MAR
Acronym: Precise MAR
Status: Not yet recruiting | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Collaborators: Philips Healthcare (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Precise MAR
Record Dates: First submitted 2025-09-23; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-09

CONDITIONS: Computed Tomography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

SUMMARY:
The purpose of this clinical study is to evaluate the performance of the P-MAR metal artifact reduction algorithm for CT imaging (with metal present) of adult patients (>18 years old).

The study has two objectives:

1. To evaluate the extent of metal artifacts and diagnostic confidence, and overall image quality (independent of metal artifacts) of P-MAR compared to images without metal correction, and compared to O-MAR, for CT images (with metal present) of adult patients (>18 years old).
2. To demonstrate non-inferiority of P-MAR compared to images without metal correction for the relevant metal groups.

ELIGIBILITY:
Inclusion Criteria:

* Subjects scanned by FDA-cleared and marketed Philips Incisive CT or CT 5300 systems, and according to the department standard of care clinical protocols.
* Subject age: Above 18 years old.
* Scans with metal present (orthopedic implants/joint prothesis, dental filling/implants, spine screw(s), pacemaker, coils, radiotherapy beads, surgical clips/staples, metal objects either outside the body or near air, etc.)

Exclusion Criteria:

* Subject age: 18 years old and below.
* CT scans with no metal present.
* CT scans with metal with motion artifacts.
* Surview or Locator/Tracker.
* CT scans performed utilizing respiratory gating (e.g., "pulmo gating").
* CT scans performed utilizing cardiac gating.
* CT Perfusion scans.
* CCT scans.
* Scans that the site radiologists have deemed as non-diagnostic image quality in standard practice (e.g. patient movement).
* Scans that are not completed due to technical difficulties.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
The extent of metal artifacts and diagnostic confidence of P-MAR | Reading session at 4 months
  The extent of metal artifacts and diagnostic confidence of P-MAR reconstructions is at least as good as (non-inferior to) images without metal correction, for CT images (with metal present) of adult patients (>18 years old).